CLINICAL TRIAL: NCT02898116
Title: A Phase 1/2 Study of ALK Inhibitor, Ensartinib (X-396), and Anti-PD-L1, Durvalumab (MEDI4736), in Subjects With ALK-rearranged (ALK-positive) Non-small Cell Lung Cancer (NSCLC)
Brief Title: Phase 1/2 Study of Ensartinib and Durvalumab, in ALK-rearranged Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: MedImmune LLC (Industry); Xcovery Holdings, Inc. (Industry); Cancer Research Institute, New York City (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUD2014-012-ALK
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Results first posted 2018-08-21 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Non-small Cell Lung Cancer; Carcinoma; NSCLC
Keywords: ALK-rearranged; ALK-positive; ALK Inhibitor; Ensartinib; X-396; anti-PD-L1; Durvalumab; MEDI4736; ALK
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma | interventions — ensartinib; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ensartinib ± Durvalumab (Experimental): Subjects were to receive ensartinib monotherapy during a pre-immunotherapy Run-in Period for one to two 28-day cycles, followed by combination therapy with ensartinib plus durvalumab for subjects with no DLTs during the Run-in Period.
  Interventions: Drug: Ensartinib; Drug: Durvalumab

INTERVENTIONS:
Drug: Ensartinib — Ensartinib was administered orally once daily at a dose of 200 mg during the Run-in Period. During combination therapy, the ensartinib starting dose was to be 200 mg. Based on observed toxicity at the starting dose level, the ensartinib dose may have been escalated to the recommended single-agent dose (225 mg) or de-escalated to the minimum effective dose (150 mg).
  Other Names: X-396
Drug: Durvalumab — During combination therapy, durvalumab was to be administered as an IV infusion over 60 (± 5) minutes every 4 weeks at a dose of 1500 mg.
  Other Names: MEDI4736

SUMMARY:
This was a Phase 1/2, open-label, multicenter, single-arm study of combination therapy with ensartinib, an anaplastic lymphoma kinase (ALK) inhibitor, and durvalumab, an anti-programmed cell death ligand 1 (PD-L1) antibody, in subjects with ALK-rearranged (ALK-positive) non-small cell lung cancer (NSCLC). Primary study objectives were to determine the recommended combination dose (RCD) and safety and tolerability of the combination. Further objectives were to evaluate the clinical efficacy and biologic activity of the combination.

DETAILED DESCRIPTION:
Prior to initiation of combination therapy with ensartinib plus durvalumab, subjects were enrolled sequentially to receive ensartinib monotherapy (orally once daily) during a pre-immunotherapy Run-in Period for one to two 28-day cycles. The purpose of the Run-in Period was to determine whether any safety signals might compromise combination therapy and to determine the effect of ALK inhibitor therapy on the immune tumor microenvironment. For subjects with no dose-limiting toxicity (DLT) during the Run-in Period, combination therapy was then initiated during a dose-finding phase using a standard 3 + 3 design until determination of the RCD, which was defined as the highest dose level at which ≤ 1 of 6 subjects (i.e., < 33%) experienced DLTs during the first 2 cycles of combination treatment.

A fixed dose of durvalumab (1500 mg by intravenous [IV] infusion every 4 weeks) was administered in all cohorts. Ensartinib dosing started at 200 mg, with subsequent cohorts receiving a reduced (150 mg) or escalated (225 mg) ensartinib dose depending upon observed toxicity. The study was then designed to include an expansion phase, in which the RCD cohort would be expanded to a total of 20 subjects.

Subjects were monitored for safety (including immune-related adverse events), disease status (using the Response Evaluation Criteria in Solid Tumors [RECIST] version 1.1 and immune-related RECIST), and biologic activity (peripheral blood assays and immunological changes in the tumor microenvironment) for the duration of study participation.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic confirmation of metastatic NSCLC. Subjects must have had confirmed ALK rearrangement as assessed by immunohistochemistry. Subjects may have had prior therapy with ALK inhibitors (other than ensartinib) or been ALK inhibitor naïve. ALK inhibitor naïve subjects were informed of the availability of approved ALK inhibitors.
2. Measurable disease according to RECIST 1.1, defined as ≥ 1 lesion that could be accurately measured in ≥ 1 dimension (longest diameter to be recorded for non-lymph node lesions, shortest diameter to be recorded for lymph node lesions). Each lesion must have been ≥ 10 mm when measured by computed tomography, magnetic resonance imaging, or caliper measurement by clinical examination or ≥ 20 mm when measured by chest x-ray.
3. Willing to provide a fresh pre-treatment biopsy; however, if subject was ALK inhibitor naïve, either archival or pre-treatment biopsy was acceptable.
4. Asymptomatic subjects with surgically treated brain metastases must have been ≥ 14 days post surgery at the time of first dosing, while clinically stable with no requirement for steroids. Asymptomatic subjects with radiation-treated brain metastases may have entered the study immediately after completion of the radiation (and been off steroids, if applicable). Symptomatic subjects (those experiencing headache, seizure etc.), must have been relieved from all symptoms of their central nervous system disease, and must have completed radiation and been off steroids prior to first dosing (anti seizure medicine permitted).
5. Laboratory parameters for vital functions should have been in the normal range. Laboratory abnormalities that were not clinically significant were generally permitted, except for the following laboratory parameters, which must have been within the ranges specified, regardless of clinical significance:

   * Hemoglobin: ≥ 9 g/dL
   * Neutrophil count: ≥ 1.5 x 10^9/L
   * Platelet count: ≥ 100,000/mm^3
   * Serum creatinine: ≤ 1.5 x institutional upper limit of normal (ULN), OR creatinine clearance: ≥ 50 mL/min (by Cockcroft-Gault formula)
   * Serum total bilirubin: ≤ 1.5 × ULN (except for subjects with Gilbert's syndrome who were allowed after consultation with their physician)
   * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT): ≤ 2.5 x ULN
   * Alkaline phosphatase: ≤ 2.5 x ULN
6. Eastern Cooperative Oncology Group Performance Status ≤ 2.
7. Age ≥ 18 years.
8. Able and willing to provide valid written informed consent.
9. Able and willing to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow-up.
10. Body weight > 30 kg.

Exclusion criteria:

1. Treatment with an investigational agent within 4 weeks of starting treatment, and any prior drug-related toxicity (except alopecia) should have recovered to Grade 1 or less.
2. Prior treatment with anti-PD-1, PD-L1 (including durvalumab), or cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4), or ensartinib (X-396).
3. Active, suspected or prior documented autoimmune disease (including but not restricted to inflammatory bowel disease, celiac disease, Wegner's granulomatosis, Hashimoto's thyroiditis, rheumatoid arthritis, systemic lupus, scleroderma and its variants, multiple sclerosis, myasthenia gravis). Vitiligo, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger were permitted.
4. Subjects with clinically significant cardiovascular disease, including:

   1. New York Heart Association Class II or higher congestive heart failure.
   2. Myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack within 6 months of start of study drug (Day -28).
   3. Clinically significant supraventricular or ventricular arrhythmia.
   4. QT interval corrected using Fridericia's formula (QTcF) ≥ 450 ms (male) or QTcF ≥ 470 ms (female).
   5. Clinically uncontrolled hypertension.
5. History of pneumonitis or interstitial lung disease, or any unresolved immune-related adverse events following prior therapy.
6. Major surgery within 4 weeks of starting treatment (or scheduled for surgery during the projected course of the study).
7. Women of child bearing potential who were pregnant as evidenced by positive serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) or nursing.
8. Female subjects of childbearing potential who were sexually active with a non-sterilized male partner must have used at least one highly effective method of contraception (see table below) from the time of screening and must have agreed to continue using such precautions for 90 days after the final dose of investigational products. Non-sterilized male partners of a female subject must have used male condoms plus spermicide throughout this period. Cessation of birth control after this point should have been discussed with a responsible physician. Not engaging in sexual activity for the total duration of the trial and the drug washout period was an acceptable practice; however, periodic abstinence, the rhythm method, and the withdrawal method were not acceptable methods of birth control.

   Female subjects should have refrained from breastfeeding throughout the period described above.

   Females of childbearing potential were defined as those who were not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or post-menopausal.

   Females were considered post-menopausal if they had been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements applied:
   * Females <50 years of age were considered post-menopausal if they had been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they had luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
   * Females ≥50 years of age were considered post-menopausal if they had been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year prior to study entry, had chemotherapy-induced menopause with last menses >1 year prior to study entry, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

   Non-sterilized male subjects who were sexually active with a female partner of childbearing potential must have used male condoms plus spermicide from screening through 90 days after receipt of the final dose of investigational products. Male subjects were to refrain from sperm donation throughout this period. Female partners (of childbearing potential) of a male subject must have used a highly effective method of contraception (see table below) throughout this period. Cessation of birth control after this point was to be discussed with a responsible physician. Not engaging in sexual activity for the total duration of the trial and the drug washout period was an acceptable practice; however, periodic abstinence, the rhythm method, and the withdrawal method were not acceptable methods of birth control.

   A highly effective method of contraception was defined as one that resulted in a low failure rate (i.e. less than 1% per year) when used consistently and correctly. Note that some contraception methods were not considered highly effective (e.g. male or female condom with or without spermicide; female cap, diaphragm, or sponge with or without spermicide; non-copper containing intrauterine device; progestogen-only oral hormonal contraceptive pills where inhibition of ovulation was not the primary mode of action [excluding Cerazette/desogestrel which was considered highly effective]; and triphasic combined oral contraceptive pills).
9. Subjects who were immunosuppressed, including those with known immunodeficiency.
10. Active infection including tuberculosis (clinical evaluation that included clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), hepatitis B (known positive hepatitis B virus surface antigen result), hepatitis C, or human immunodeficiency virus (positive 1/2 antibodies). Subjects with a past or resolved hepatitis B virus infection (defined as the presence of hepatitis B core antibody and absence of hepatitis B virus surface antigen) were eligible. Subjects positive for hepatitis C antibody were eligible only if polymerase chain reaction was negative for hepatitis C virus ribonucleic acid.
11. History of severe allergic reactions to any unknown allergens or components of the study drugs.
12. Other serious illnesses (e.g., serious infections requiring antibiotics, bleeding disorders).
13. Mental impairment that may have compromised compliance with the requirements of the study.
14. Lack of availability for immunological and clinical follow-up assessment.
15. Inability to swallow or retain oral medication, presence of active gastrointestinal disease or other condition that would have interfered significantly with the absorption, distribution, metabolism, or excretion of ensartinib.
16. Any condition that, in the clinical judgment of the treating physician, was likely to prevent the subject from complying with any aspect of the protocol or that may have put the subject at unacceptable risk.
17. History of allogeneic organ transplant.
18. Subjects must not have donated blood while on study and for at least 90 days following the last durvalumab treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2017-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leena Gandhi, MD, PhD, Study Chair — Laura & Isaac Perlmutter Cancer Center
Locations (1):
- Research Facility, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ensartinib (200 mg): Subjects received ensartinib monotherapy (200 mg orally once daily) during a pre-immunotherapy Run-in Period for one to two 28-day cycles.
Period: Overall Study
Arm/Group | Ensartinib (200 mg)
Started | 2
Completed | 0
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Progressive disease | 1

BASELINE CHARACTERISTICS:
Population: All enrolled subjects
Arm/Group | Ensartinib (200 mg)
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 57 [48 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-emergent Adverse Events
Description: Toxicity was graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.03. Treatment-emergent adverse events (TEAEs) were reported based on clinical laboratory tests, physical examinations, and vital signs from pre-treatment through the end of the study period. Dose-limiting toxicity (DLT) during the Run-in Period was defined as ≥ Grade 2 rash or other toxicity requiring discontinuation of ensartinib dosing.
Time Frame: up to 3 months
Population: All enrolled subjects
Measure: Number; unit: participants
Arm/Group | Ensartinib (200 mg)
Number analyzed (Participants) | 2
participants
  Any TEAE | 2
  Maximum grade 2 TEAE | 1
  Maximum grade 3 TEAE | 1
  Immune-related TEAE | 0
  Ensartinib-related TEAE | 2
  Serious TEAE | 1
  TEAE Leading to Discontinuation | 1
  TEAE Meeting DLT Criteria | 0

2. Secondary Outcome: Number of Subjects With Best Overall Tumor Response at the Last Assessment
Description: Tumor response was evaluated using computed tomography and categorized according to the Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1) at Baseline, every 2 cycles, and at the end of the study. Per RECIST, target lesions are categorized as follows: Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; Stable Disease (SD): small changes that do not meet above criteria.
Time Frame: up to 3 months
Population: All enrolled subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Ensartinib (200 mg)
Number analyzed (Participants) | 2
Participants
  SD | 0
  PD | 2

3. Secondary Outcome: Number of Subjects With Immune-related Tumor Response at the Last Assessment
Description: Immune-related tumor response was evaluated by computed tomography at Baseline, every 2 cycles, and at the end of the study. Tumor response was designated according to the immune-related Response Criteria (irRC) (Wolchok et al. Clin Cancer Res 2009;15:7412-20) into the following categories: immune-related complete response (irCR) requires disappearance of all lesions in two consecutive observations not less than 4 weeks apart; immune-related partial response (irPR) requires ≥ 50% decrease in tumor burden compared with baseline in two observations at least 4 weeks apart; immune-related stable disease (irSD) is assigned when neither a 50% decrease from baseline tumor burden nor a 25% increase in tumor burden from nadir can be established; immune-related progressive disease (irPD) requires a ≥ 25% increase from nadir in tumor burden at any single time point in two consecutive observations at least 4 weeks apart.
Time Frame: up to 3 months
Population: All enrolled subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Ensartinib (200 mg)
Number analyzed (Participants) | 2
Participants
  irSD | 0
  irPD | 2

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) occurring between the signing of informed consent and the off-study date were documented, regardless of the causal relationship to study drug. AEs occurring after the first dose of study drug were considered treatment emergent (i.e., TEAEs). The AE reporting period for this study was up to 3 months.
Description: AE documentation included onset/resolution dates, severity using the NCI CTCAE (version 4.03), seriousness, relationship to study drug, study drug action taken, treatment, and outcome. In summaries, treatment-related AEs included those with a "possible", "probable", or "definite" relationship to study drug; preferred terms were counted only once per subject at the maximum reported grade.
Arm/Group | Ensartinib (200 mg)
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ensartinib (200 mg) (N=2)
Hypersensitivity (Immune system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ensartinib (200 mg) (N=2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pyrexia (General disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Eosinophilia (Blood and lymphatic system disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Blood alkaline phosphatase increased (Investigations) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Insomnia (Psychiatric disorders) | 1
Fatigue (General disorders) | 1
Weight decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Nausea (Gastrointestinal disorders) | 1

LIMITATIONS AND CAVEATS:
Early termination due to the rapidly changing treatment landscape for ALK-positive NSCLC, resulting in low enrollment. Because only 2 subjects were enrolled, no separate statistical analysis plan was issued and no formal data analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT02898116/Prot_SAP_000.pdf